CLINICAL TRIAL: NCT00443807
Title: A Comparison of the EEGo and BIS Monitors to Assess Emergence From Neuroanesthesia
Brief Title: EEG Monitoring to Assess Emergence From Neuroanesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: W. Alan C. Mutch, University of Manitoba
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: B2007:008
Record Dates: First submitted 2007-03-05; First posted 2007-03-06 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-04

CONDITIONS: Cerebral Aneurysm; Trigeminal Neuralgia
MeSH Terms: conditions — Intracranial Aneurysm; Trigeminal Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: On-line EEG monitoring during neurosurgery — Comparison of 2 ways of processing the EEG signal
  Other Names: EEGo; BIS Vista
Device: EEGo vs BIS — comparison of two processed EEG monitors.

SUMMARY:
A highly desired result in neuroanesthesia is a prompt, controlled emergence following a neurosurgical procedure. Considerable strides have been made in this direction with volatile anesthetic agents such as sevoflurane or desflurane administered in association with the narcotic remifentanil. It is characteristic that patients will emerge within 5 to 10 minutes of cessation of these agents at the end of a neuroanesthetic. However, there are cases where emergence is delayed, especially after periods of deep anesthesia for i) cerebral protection with temporary clipping of cerebral aneurysms and ii) with microvascular decompression for trigeminal neuralgia. Deep levels of anesthesia are standard for these procedures in the posterior fossa, which utilize motor evoked potentials to assess cranial nerve function. In these cases, EEG monitoring is standard. Using the EEG to monitor emergence to aid its progress makes sense. A monitor which could predict emergence in these patients would be valuable. EEG monitoring engineered to provide this information is now available in the form of the EEGo. This study is designed to test the hypothesis that the EEGo monitor will be superior to the BIS monitor to assess emergence following neuroanesthesia.

DETAILED DESCRIPTION:
Objective: This study is designed to test the hypothesis that the EEGo monitor will be superior to the BIS monitor to assess emergence following neuroanesthesia. The EEGo will be able to more accurately indicate emergence and direct therapy at the end of the operative procedure. The EEGo will be superior because the raw EEG signal is processed using phase delay analysis, with each patient's raw EEG analyzed instead of a proprietary but generic signal processing approach on a linear scale as with the BIS monitor. Phase delay analysis is a standard approach to display nonlinear signals. A highly reproducible signal transition occurs from deep anesthesia to emergence. It is this transition that permits acute assessment of emergence. The ability to process the EEG and display phase delay plots in 50 msec is what makes the EEGo monitor attractive to acutely assess emergence from neuroanesthesia. Accurate emergence will allow better anesthesia management.

This pilot study will be done to assess a nonlinear EEG monitor (EEGo) to direct therapy and predict prompt emergence from neuroanesthesia where EEG monitoring is done in neurosurgical cases. In our centre we routinely monitor the EEG, SSEP and/or MEP during temporary aneurysm clipping and during microvascular decompressive surgery. It is just these cases where emergence can be delayed despite following standard neuroanesthesia techniques. The EEGo processes the standard EEG signal by nonlinear analysis of the raw signal by 3 dimensional phase delay plots. A cascade from a point attractor, periodic attractor, toroidal attractor to a 3-D chaotic attractor occurs from burst suppression to the awake state. These resemble phase transitions and occur rapidly from one state to the next. An analogy is the phase transition that occurs when water changes to ice and vice versa. Monitoring these transitions should permit a rational approach to therapy during anesthesia emergence, better predict emergence, facilitate extubation based on the awake state, allow titration of vasoactive agents during emergence to smooth hemodynamic control and permit more rapid emergence at end procedure. The EEGo will be compared directly in real time to the bispectral (BIS) monitor re goal directed emergence. If efficacy is shown with the EEGo, a more formal comparison to BIS and clinical judgement will be studied.

BIS monitoring can aid emergence in outpatient procedures, both with time to wakening and time in the recovery room. These results also impact on the cost of anesthetic drugs and OR and Recovery Room costs. Work demonstrating accelerated emergence from desflurane with BIS do not highlight the manner in which the BIS directs the emergence. The depth of anesthesia is adjusted to 50 - 60 ABU during maintenance and then emergence is tracked. A specific BIS number to indicate emergence is not suggested. In fact, a correlation between the BIS in the awake state and with movement and eye opening appears poor with the emergence BIS usually being lower than the pre-induction BIS. The BIS may also on occasion be very low during emergence - deemed artifactually so and in this work it is suggested that the raw EEG be observed to aid emergence. It would seem that significant issues relate to intra and interpatient variability with this processed EEG signal. Recent work suggests significant discrepancy of BIS signals between hemispheres and even recording from two sites in the same hemisphere. In addition, BIS correlates poorly with end-tidal desflurane and awake state.

Thus, it would seem that while the BIS can aid management of depth of anesthesia during maintenance, it is not ideally suited to direct a facilitated emergence. In contrast, the EEGo monitor uses nonlinear analysis techniques to provide a visual output related to depth of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing neurosurgery where intraoperative EEG monitoring is the standard of care will be approached in the Pre-Anesthetic Clinic for participation.

Exclusion Criteria:

* Patient refusal
* a history of asthma requiring routine use of bronchodilators, because the study will use desflurane as the volatile agent
* pregnancy
* non-elective aneurysm clipping

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
An assessment of quality of emergence - smooth, single cough, multiple coughs will be provided by the neurosurgeon | Wake up time in OR

SECONDARY OUTCOMES:
Twenty-four hours post surgery a directed survey of patient satisfaction and questioning regarding awareness will be done | hours

CONTACTS AND LOCATIONS:
Overall Officials: W. Alan C. Mutch, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada